CLINICAL TRIAL: NCT03887468
Title: Dialysis Adequacy and Clotting Complications During Anticoagulation-free Hemodialysis Using a Heparin-grafted Dialyzer and a Citrate-enriched Dialysate: a Prospective Randomized Crossover Study. (EvoCit-HD Study)
Brief Title: Hemodialysis Adequacy Using a Heparin-grafted Dialyzer and a Citrate-enriched Dialysate
Acronym: EvoCit-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UZB-NEF-2017-EvoCit-HD
Record Dates: First submitted 2019-01-22; First posted 2019-03-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Kidney Diseases; Hemodialysis Complication; End Stage Renal Disease
Keywords: dialysis adequacy; clotting
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "EvoCit" (Active Comparator): Standardized hemodialysis treatments 3x4hours/week. Intervention: "EvoCit procedure" using a heparin-grafted AN69ST dialyzer in combination with a citric acid enriched dialysate without any systemic anticoagulation.
  Interventions: Device: EvoCit
- "EvoHep" (Active Comparator): Control: "EvoHep procedure" using a heparin-grafted AN69ST dialyzer in combination with a conventional bicarbonate-based dialysate and standardized systemic anticoagulation using unfractionated heparin.
  Interventions: Device: EvoHep

INTERVENTIONS:
Device: EvoCit — hemodialysis using the combination of the Evodial dialyzer with a citrate enriched dialysate
  Arms: "EvoCit"
Device: EvoHep — hemodialysis using the combination of the Evodial dialyzer with a conventional bicarbonate based dialysate and systemic anticoagulation using unfractionated heparin
  Arms: "EvoHep"

SUMMARY:
After providing informed consent, patients will be randomized to either the intervention treatment ("EvoCit procedure") or the control treatment ("EvoHep procedure").

After randomization, each study arm consists of four weeks of 3x4 hours hemodialysis treatments according to the allocated protocol. After the last dialysis treatment of the fourth treatment week and after a long interdialytic interval, patients will crossover to the alternative hemodialysis procedure. After crossover, the study will be completed with, again, four weeks of 3x4 hours hemodialysis treatments according to the allocated protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with hemodialysis or hemodiafiltration since at least three months.
* Hemodialysis or hemodiafiltration prescription of 3 x 4 hours weekly.
* ≥ 18 years of age.
* Patients able and agree to provide signed informed consent.

Exclusion Criteria:

* Contraindication to heparin defined as known heparin-induced thrombopenia or active bleeding risk with contra-indication for systemic anticoagulation, categorized as defined by Swartz and Port1.
* Planned surgery during study period, including scheduled living-donor kidney transplantation during study period.
* Hypercoagulable state defined as known malignancy, known APC resistance/FV Leiden, known prothrombin gene mutation, known protein C or protein S deficiency, known antithrombin deficiency.
* Mean Qb of <300ml/min during one of the last 3 dialysis sessions before inclusion.
* 1 or more results of spKt/Vurea < 1,35 during the last three months prior to study inclusion.
* Need for 2 or more supplementary dialysis sessions on top of the regular 3x4 hours weekly hemodialysis regimen during the last month before inclusion.
* Vascular access dysfunction defined as

  1. use of urokinase the 2 months before study inclusion, including to restore catheter permeability.
  2. non-tunneled hemodialysis catheter use.
  3. known AV access outflow tract stenosis.
  4. planned vascular access intervention.
  5. planned vascular access conversion.
* Known allergy against heparin grafted AN69STmembranes.
* Use of ACE-inhibitor
* Use of vitamin K antagonist
* Use of novel oral anticoagulant therapy.
* Any medical condition, which puts the patient at risk of premature study termination in the opinion of the investigator.
* Planned conversion of dialysis modality during study period or planned absence/leave (including pregnancy or planned pregnancy).
* Symptomatic hypocalcemia.
* Hb < 8g/dl at screening.
* Hct > 45% at screening.
* Perdialytic total parenteral nutrition therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
change in dialysis adequacy | every midweek dialysis session through study duration, ie 2x4 weeks
  spKt/Vurea

SECONDARY OUTCOMES:
proportion of thrombotic dysfunction | every HD session through study duration, ie 2x4 weeks
  premature termination of the dialysis session
change in dialysis adequacy expressed by middle molecule (MM) clearance | every 1st and 4th week HD session through study duration, ie 2x4 weeks
  MM clearances
occurence of complete circuit thrombosis | every HD session through study duration, ie 2x4 weeks
  rapidly occurring thrombosis of the extracorporeal circuit, which does not allow complete retransfusion of the blood circuit even if prescribed treatment duration is reached
change in membrane coagulation | every midweek HD session through study duration, ie 2x4 weeks
  total cell volume measurement of the dialyzer after hemodialysis
occurence of biological evaluation of coagulation activation | every 1st and 4th week HD session through study duration, ie 2x4 weeks
  TAT, PF1+2,

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette
  - CHU Brugmann, Laken

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Francois K, De Clerck D, Tonnelier A, Cambier ML, Orlando C, Jochmans K, Cools W, Wissing KM. Dialyzer Performance During Hemodialysis Without Systemic Anticoagulation Using a Heparin-Grafted Dialyzer Combined With a Citrate-Enriched Dialysate: Results of the Randomized Crossover Noninferiority EvoCit Study. Am J Kidney Dis. 2022 Jan;79(1):79-87.e1. doi: 10.1053/j.ajkd.2021.04.004. Epub 2021 Apr 30. PMID 33940113